CLINICAL TRIAL: NCT00232622
Title: A Prospective Randomized Trial of a Rapid Fibrinolytic Protocol for Left-sided Prosthetic Valve Thrombosis
Brief Title: A Study Comparing a New Dosing Regimen of Clot-dissolving Drug for Mechanical Heart Valves Which Show Clots
Acronym: RAFT-PVT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Ganesan Karthikeyan, Additional Professor of Cardiology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-29/3.3.2004
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Prosthetic Valve Thrombosis
Keywords: Prosthetic valve thrombosis; Fibrinolysis; Streptokinase
MeSH Terms: interventions — Streptokinase; Thrombolytic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard infusion of streptokinase (Active Comparator): Standard infusion of streptokinase
  Interventions: Drug: Streptokinase
- Accelerated infusion of streptokinase (Experimental): Accelerated infusion of streptokinase
  Interventions: Drug: Streptokinase

INTERVENTIONS:
Drug: Streptokinase — Accelerated infusion of streptokinase
  Other Names: Fibrinolytic therapy
  Arms: Accelerated infusion of streptokinase
Drug: Streptokinase — Standard dose streptokinase
  Other Names: Fibrinolytic therapy
  Arms: Standard infusion of streptokinase

SUMMARY:
The optimal dosage and duration of administration of clot-dissolving medications for the treatment of patients with mechanical heart valves with clots is not known. We hypothesized that a large dose of the clot-dissolving medicine given initially (akin to the dose given in the treatment of heart attacks), might speed up the dissolution of the clot and rapidly restore the functioning of the mechanical heart valve.

DETAILED DESCRIPTION:
The optimal fibrinolytic strategy for left sided prosthetic valve thrombosis (PVT) is not known. A large initial bolus dose of streptokinase (SK) might accelerate fibrinolysis and restore valve function more rapidly.

This is a prospective, randomized trial comparing 2 fibrinolytic protocols in a first episode of PVT. In the rapid fibrinolytic protocol (RFP) 1.5 MU of SK is given over 1 hour, followed if required by a 0.1 MU/h infusion. In the standard protocol (SP) 0.25 MU is given over 30 minutes, followed by an infusion of 0.1 MU/h. Serial echocardiography and fluoroscopy will be done to monitor therapy. The primary end point is the occurrence of a complete clinical response (CCR, complete hemodynamic response without any major complication). 58 patients are required in each arm for detecting a 30% difference with 80% power at α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* First episode of left sided prosthetic valve thrombosis

Exclusion Criteria:

* Contraindication to thrombolysis
* Refusal to give informed consent
* Pregnant women
* age less than 12 years or more than 70 years
* previous treatment for prosthetic valve thrombosis

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The occurrence of a complete clinical response (complete hemodynamic response as assessed by echocardiography and fluoroscopy, without any major complication) | In-hospital

SECONDARY OUTCOMES:
Death, Major bleeding and minor bleeding | In-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ganesan Karthikeyan, MD, DM, Principal Investigator — Department of Cardiology, All India Institute of Medical Sciences

REFERENCES:
- [Result] Karthikeyan G, Math RS, Mathew N, Shankar B, Kalaivani M, Singh S, Bahl VK, Hirsh J, Eikelboom JW. Accelerated infusion of streptokinase for the treatment of left-sided prosthetic valve thrombosis: a randomized controlled trial. Circulation. 2009 Sep 22;120(12):1108-14. doi: 10.1161/CIRCULATIONAHA.109.876706. Epub 2009 Sep 8. PMID 19738134
- [Result] Karthikeyan G, Mathew N, Math RS, Devasenapathy N, Kothari SS, Bahl VK. Timing of adverse events during fibrinolytic therapy with streptokinase for left-sided prosthetic valve thrombosis. J Thromb Thrombolysis. 2011 Aug;32(2):146-9. doi: 10.1007/s11239-011-0579-4. PMID 21416132
- [Derived] Barwad P, Raheja A, Venkat R, Kothari SS, Bahl V, Karthikeyan G. High prevalence of silent brain infarction in patients presenting with mechanical heart valve thrombosis. Am J Cardiovasc Drugs. 2012 Oct 1;12(5):345-8. doi: 10.1007/BF03261843. PMID 22779430